CLINICAL TRIAL: NCT06784336
Title: Phase II Multi-center Study of Resistant Potato Starch Plus Deferasirox to Improve Outcomes in Patients Undergoing Allogeneic Stem Cell Transplantation
Brief Title: Phase II Study of Resistant Potato Starch Plus Deferasirox to Improve Outcomes in Patients Undergoing Allogeneic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2024.092; HUM00262804 (Other: University of Michigan)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Allogeneic Stem Cell Transplant
MeSH Terms: interventions — Iron Chelating Agents; Deferasirox

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Treatment (Experimental): All subjects will be enrolled into one arm and will be treated with RPS and Iron Chelation
  Interventions: Drug: Iron chelation; Drug: Potato Resistant Starch

INTERVENTIONS:
Drug: Iron chelation — Patients will receive Iron chelation with deferasirox (Jadenu 7 mg/kg/day preferred versus Exjade 10 mg/kg/day) beginning on day -14 and continuing through day +100
  Other Names: Deferasirox
Drug: Potato Resistant Starch — Patients will receive PRS beginning on day -6 and continuing through day +100. Patients will take 20g packet twice daily
  Other Names: Bob's Red Mill

SUMMARY:
The study will evaluate the safety and early efficacy of administering the combination of a commercially available potato-based resistant starch along with iron chelation therapy to subjects undergoing alloHCT.

DETAILED DESCRIPTION:
The deferasirox intervention will begin one week prior to the RPS (Resistant Potato Starch) conditioning phase and both will continue through day +100. The study hypothesis is that a short-term administration of a resistant starch and iron chelation therapy will be capable of both increasing levels of butyrate within the intestine and restoring physiological hypoxia in the intestines, which together will reduce rates of acute GVHD (Graft versus Host Disease) and improve the clinically meaningful outcome of GRFS (Graft versus Host Disease / Relapse-Free Survival) at 12 months post-transplant.

21NOV2025- The grant previously listed on this trial is associated with the conduct of a preliminary study NCT02763033. Therefore, it was removed from this clinical trial as it is not being used for the conduct of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic disorders undergoing allo-HCT from fully HLA-matched unrelated or related donors after full-intensity conditioning regimen
* Age ≥18 years
* Karnofsky performance status >70%, see Appendix A
* Patients must be able to swallow capsules/tablets
* Ability to understand and the willingness to sign a written informed consent
* Availability of a full-HLA matched related or unrelated donor who is medically eligible to donate cells according to the National Marrow Donor Program criteria

Exclusion Criteria:

* Patients with active inflammatory bowel disease requiring treatment per treating investigator
* Patients with a history of gastric bypass surgery
* Patients with active Clostridium difficile infection at the time of study enrollment. Active infection is defined as a stool sample positive for Clostridium difficile toxin via enzyme immunoassay (EIA) and either symptoms (frequent loose stools) OR imaging findings consistent with toxic megacolon
* Patients with active iron deficiency anemia requiring treatment
* Patients with iron overload receiving active treatment with deferasirox
* Known hypersensitivity to deferasirox or any component of Jadenu or Exjade
* Patients actively enrolled on treatment or in follow up phase on any other GVHD prevention trial
* Any physical or psychological condition that, in the opinion of the investigator, would pose an unacceptable risk to the patient or raise concern that the patient would not comply with protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
GVHD-free and relapse-free survival | up to 1 year post- transplantation
  Assessed in a time-to-event analysis, with GRFS defined as the first occurrence of grade III or IV acute GVHD, chronic GVHD warranting systemic immunosuppression, disease relapse or progression, or death from any cause.

SECONDARY OUTCOMES:
Rates of grade II, III and IV acute GVHD | up to 1 year post- transplantation
  Cumulative incidence of grades II to IV GVHD and of grades III to IV acute GVHD
Rates of chronic GVHD requiring systemic immunosuppression | up to 1 year post- transplantation
  Cumulative incidence of chronic GVHD warranting systemic immunosuppression
Length of event-free survival | up to 1 year post- transplantation
  time to relapse/progression or death as first event

CONTACTS AND LOCATIONS:
Overall Officials: Mary Riwes, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No